CLINICAL TRIAL: NCT00596271
Title: Safety and Immunogenicity of Concomitant Vaccination With IC51 and HARVIX® 1440 in Healthy Subjects. A Single-blind Randomized, Controlled Phase 3 Study
Brief Title: Concomitant Vaccination With the Japanese Encephalitis Vaccine IC51 and HARVIX® 1440
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IC51-308
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Results first posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-04

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese | interventions — Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- IC51 and Placebo (Active Comparator): 6 mcg i.m. IC51 with 2 injections (day 0 and 28)and placebo 0.5 mL with 1 injection (day 0)
  Interventions: Biological: IC51; Other: Placebo
- HAVRIX and placebo (Active Comparator): HAVRIX with 1 injection (day 0) and placebo 0.5 mL with 2 injections (day 0 and 28)
  Interventions: Biological: HAVRIX; Other: Placebo
- IC51 and HAVRIX (Active Comparator): IC51 6 mcg i.m. with 2 injections (day 0 and 28) and HAVRIX with 1 injection (day 0)
  Interventions: Biological: IC51; Biological: HAVRIX

INTERVENTIONS:
Biological: IC51
  Other Names: Japanese Encephalitis purified inactivated vaccine
  Arms: IC51 and HAVRIX; IC51 and Placebo
Biological: HAVRIX
  Arms: HAVRIX and placebo; IC51 and HAVRIX
Other: Placebo
  Arms: HAVRIX and placebo; IC51 and Placebo

SUMMARY:
The objective is to investigate the immunogenicity of the Japanese Encephalitis vaccine IC51 (JE-PIV) single and concomitant with HAVRIX® 1440

DETAILED DESCRIPTION:
This is a randomized, controlled, multi-center, single-blind phase 3 study. The study population consists of male and female healthy subjects, aged at least 18 years.

192 subjects will be enrolled at 2 sites in Europe.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* In female subjects either childbearing potential terminated by surgery or one year post-menopausal, or a negative serum pregnancy test during screening and the willingness not to become pregnant during the study period and 30 days after the last vaccination by practicing reliable methods of contraception
* Written informed consent obtained prior to study entry

Exclusion Criteria:

* History of clinical manifestation of any flavivirus infection
* History of vaccination against Japanese encephalitis (JE), Yellow fever and Dengue fever (an anti-JEV neutralizing antibody titer >= 1:10 at baseline is acceptable for inclusion, these subjects will be part of the safety population, but will not be analyzed for immunogenicity in the per-protocol analysis)
* History of any previous Hepatitis A vaccination and infection
* Use of any other investigational or non-registered drug or vaccine in addition to the study vaccine during the study period or within 30 days preceding the first dose of study vaccine
* Planned administration of another vaccine during the study period
* Immunodeficiency including post-organ-transplantation or immunosuppressive therapy
* A family history of congenital or hereditary immunodeficiency
* History of autoimmune disease
* Administration of chronic (defined as more than 14 days) immunosuppressants or other immune-modifying drugs within six months of vaccination.
* Any acute infections within 4 weeks prior to enrollment
* Infection with human immunodeficiency virus (HIV), Hepatitis B (HBsAg) or Hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2005-09; Primary Completion 2006-07 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Kaltenboeck, Ph.D., Study Director — Valneva Austria GmbH

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject In: 26.09.2005, Last Subject Out: 14.07.2006 performed at centers for travelling medicine/vaccinology
Period: Overall Study
Arm/Group | IC51 and Placebo | HAVRIX and Placebo | IC51 and HAVRIX
Started | 65 | 65 | 62
Completed | 60 | 59 | 61
Not Completed | 5 | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IC51 and Placebo | HAVRIX and Placebo | IC51 and HAVRIX | Total
Number analyzed (Participants) | 65 | 65 | 62 | 192
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 65 | 65 | 62 | 192
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 35 | 34 | 103
  Male | 31 | 30 | 28 | 89
Region of Enrollment [Number; unit: participants]
  Europe | 65 | 65 | 62 | 192

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) at Day 56 for Anti-JEV Neutralizing Antibodies
Description: anti-JEV Neutralizing Antibodies were tabulated for IC51 groups only; for HAV GMTs (co-primary endpoint GMT for Hepatitis A Virus (HAV) Antibody at Day 28), please refer to "Outcome 2" within outcome measure section
Time Frame: Day 56
Population: Per Protocol Population includes all randomized subjects without major protocol deviations
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | IC51 and Placebo | IC51 and HAVRIX
Number analyzed (Participants) | 58 | 58
titers | 192.2 [147.9 to 249.8] | 202.7 [153.7 to 261.2]
Statistical Analysis 1: Comparison: IC51 and Placebo vs IC51 and HAVRIX; The primary efficacy analysis will compare the IC51+HAVRIX vs. IC51+Placebo group in terms of the GMT for anti- JEV neutralizing antibody at day 56. An observed cases approach will be applied for the primary analysis; Test type: Non-Inferiority or Equivalence — Non-inferiority of the combined administration is postulated, if the lower bounds of both twosided 95% confidence intervals for the GMT ratios (of combined vaccination over single vaccination) are > 1/2. This procedure is equivalent to the approach based on a 1-sided test with a significance level of 2.5% for each comparison with the null hypothesis H0 : ratio ≤ 0.5 versus the alternative hypotheses H1 : ratio > 0.5; p < 0.0001, ANOVA

2. Secondary Outcome: Seroconversion Rate (SCR) at Day 56 for Plaque Reduction Neutralization Assay (PRNT) and HAV at Day 28
Time Frame: day 28 and 56
Reporting Status: Not Posted

3. Secondary Outcome: GMT and SCR for PRNT at Day 28 and HAV at Day 56
Time Frame: day 28 and 56
Reporting Status: Not Posted

4. Secondary Outcome: Safety
Description: Rate of Adverse Events (AEs), Serious Adverse Events (SAEs) and medically attended AEs, local and systemic tolerability, changes in safety laboratory parameters (hematology, serum chemistry, urinalysis)
Time Frame: until 6 month after last vaccination
Reporting Status: Not Posted

5. Primary Outcome: GMT for Hepatitis A Virus (HAV) Antibody at Day 28
Time Frame: Day 28
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | HAVRIX + Placebo | IC51 + HAVRIX
Number analyzed (Participants) | 52 | 58
titers | 21.7 [17.2 to 27.5] | 24 [19.1 to 30.1]
Statistical Analysis 1: Comparison: HAVRIX + Placebo vs IC51 + HAVRIX; The primary efficacy analysis will compare the IC51+HAVRIX vs. HAVRIX+Placebo group in terms of the GMT for HAV antibody at day 28. An observed cases approach will be applied for the primary analysis; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA

ADVERSE EVENTS:
Arm/Group | IC51 and Placebo | HAVRIX and Placebo | IC51 and HAVRIX
Serious Adverse Events (participants affected / at risk) | 1/65 | 0/65 | 0/62
Other Adverse Events (participants affected / at risk) | 27/65 | 31/65 | 24/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IC51 and Placebo (N=65) | HAVRIX and Placebo (N=65) | IC51 and HAVRIX (N=62)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IC51 and Placebo (N=65) | HAVRIX and Placebo (N=65) | IC51 and HAVRIX (N=62)
Fatique (General disorders) | 2 | 5 | 5
Influenza like illness (General disorders) | 6 | 3 | 3
Pyrexia (General disorders) | 2 | 0 | 2
Nasopharyngitis (Infections and infestations) | 4 | 4 | 5
Cystitis (Infections and infestations) | 1 | 1 | 2
Rhinitis (Infections and infestations) | 2 | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 2
Gastrointeritis (Infections and infestations) | 0 | 1 | 2
Rash pustular (Infections and infestations) | 0 | 2 | 0
Headache (Nervous system disorders) | 4 | 10 | 4
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 4
Nausea (Gastrointestinal disorders) | 2 | 2 | 2
Hepatic enzyme increased (Investigations) | 2 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other